CLINICAL TRIAL: NCT03054428
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Dupilumab Monotherapy in Patients ≥12 to <18 Years of Age, With Moderate-to-severe Atopic Dermatitis
Brief Title: Efficacy and Safety of Dupilumab in Participants ≥12 to <18 Years of Age, With Moderate-to-severe Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-AD-1526; 2015-004458-16 (EudraCT Number)
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Moderate-to-Severe Atopic Dermatitis; Dermatitis, Dermatitis Atopic; Eczema, Skin Diseases, Skin; Diseases Genetic, Genetic; Diseases Inborn, Skin; Disease, Eczematous Skin; Hypersensitivity, Immediate; Hypersensitivity, Immune System Diseases; Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Skin Diseases; Genetic Diseases, Inborn; Skin Diseases, Eczematous; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Experimental): Participants received placebo matching dupilumab once every 2 weeks (Q2W) (including doubling the amount of placebo on day 1 to match the loading dose). In order to maintain blinding for the study, participants in the <60 kilogram (kg) weight stratum received, in a 1:1 ratio, either placebo matching 200 milligram (mg) dupilumab (including doubling the amount of placebo on day 1 to match the loading dose) or placebo matching 300 milligram (mg) dupilumab (including doubling the amount of placebo on day 1 to match the loading dose). In the ≥60 kg weight stratum, the participants randomized to the placebo group received placebo matching 300 mg dupilumab (including doubling the amount of placebo on day 1 to match the loading dose).
  Interventions: Drug: Placebo
- Dupilumab 300 mg Q4W (Experimental): Participants received once every 4 weeks (Q4W) subcutaneous (SC) injections of 300 milligrams (mg) dupilumab following a loading dose of 600 mg on day 1. In order to maintain blinding, all participants received an injection once every 2 weeks (Q2W) from day 1 to week 14. Participants received placebo 2 milliliter (mL) injection at the weeks dupilumab was not given.
  Interventions: Drug: Dupilumab
- Dupilumab 200 mg or 300 mg Q2W (Experimental): Participants with baseline weight <60 kg received once every 2 weeks (Q2W) subcutaneous (SC) injections of 200 milligrams (mg) dupilumab following a loading dose of 400 mg on day 1. Participants with baseline weight ≥60 kg received Q2W SC injections of 300 mg dupilumab following a loading dose of 600 mg on day 1.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Subcutaneous injection among the different quadrants of the abdomen (avoiding navel and waist areas), upper thighs, and upper arms.
  Other Names: REGN668
  Arms: Dupilumab 200 mg or 300 mg Q2W; Dupilumab 300 mg Q4W
Drug: Placebo — Subcutaneous injection among the different quadrants of the abdomen (avoiding navel and waist areas), upper thighs, and upper arms.
  Arms: Placebo

SUMMARY:
The primary objective of the study was to demonstrate the efficacy of dupilumab as a monotherapy in participants ≥12 years to <18 years of age with moderate-to-severe atopic dermatitis (AD). The secondary objective of the study was to assess the safety of dupilumab as a monotherapy in participants ≥12 years to <18 years of age with moderate-to-severe AD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥12 to <18 years of age at time of screening visit
* Diagnosis of AD according to the American Academy of Dermatology consensus criteria at screening visit
* IGA ≥3 at screening and baseline visit
* EASI ≥16 at the screening and baseline visit
* Baseline Pruritus NRS average score for maximum itch intensity ≥4
* ≥10% BSA of AD involvement at the screening and baseline visits
* With documented recent history (within 6 months before the screening visit) of inadequate response to topical AD medication(s) or for whom topical treatments is medically inadvisable

Exclusion Criteria:

* Participation in a prior dupilumab clinical study
* Treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within 2 weeks before the baseline visit
* Having used immunosuppressive/immunomodulating drugs within 4 weeks before the baseline visit
* Body weight <30 kg at baseline
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiprotozoals, or antifungals within 2 weeks before the baseline visit
* Known or suspected immunodeficiency, known history of human immunodeficiency virus (HIV) infection or HIV seropositivity at the screening visit, established diagnosis of HBV infection or HBV seropositivity at screening, established diagnosis of HCV infection or HCV seropositivity at screening
* History of malignancy before the baseline visit
* Diagnosed active endoparasitic infections or at high risk of these infections
* Patient is female who is pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study
* Patient is female of childbearing potential and sexually active, who is unwilling to use adequate methods of contraception throughout the duration of the study and for 120 days after the last dose of study drug

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (42):
- United States (34):
  - Regeneron Investigational Site, Birmingham, Alabama
  - Regeneron Investigational Site, Gilbert, Arizona
  - Regeneron Investigational Site, Bakersfield, California
  - Regeneron Investigational Site, Long Beach, California
  - Regeneron Investigational Site, Rolling Hills Estates, California
  - Regeneron Investigational Site, San Diego, California
  - Regeneron Investigational Site, Santa Rosa, California
  - Regeneron Investigational Site, Centennial, Colorado
  - Regeneron Investigational Site, Denver, Colorado
  - Regeneron Investigational Site, Washington D.C., District of Columbia
  - Regeneron Investigational Site, Tampa, Florida
  - Regeneron Investigational Site, Macon, Georgia
  - Regeneron Investigational Site, Sandy Springs, Georgia
  - Regeneron Investigational Site, Chicago, Illinois
  - Regeneron Investigational Site, Evansville, Indiana
  - Regeneron Investigational Site, Indianapolis, Indiana
  - Regeneron Investigational Site, Plainfield, Indiana
  - Regeneron Investigational Site, Rockville, Maryland
  - Regeneron Investigational Site, Boston, Massachusetts
  - Regeneron Investigational Site, Plymouth, Minnesota
  - Regeneron Investigational Site, St Louis, Missouri
  - Regeneron Investigational Site, Forest Hills, New York
  - Regeneron Investigational Site, New York, New York
  - Regeneron Investigational Site, Rochester, New York
  - Regeneron Investigational Site, Chapel Hill, North Carolina
  - Regeneron Investigational Site, Bexley, Ohio
  - Regeneron Investigational Site, Tulsa, Oklahoma
  - Regeneron Investigational Site, Portland, Oregon
  - Regeneron Investigational Site, Philadelphia, Pennsylvania
  - Regeneron Investigational Site, Charleston, South Carolina
  - Regeneron Investigational Site, Bellaire, Texas
  - Regeneron Investigational Site, San Antonio, Texas
  - Regeneron Investigational Site, Norfolk, Virginia
  - Regeneron Investigational Site, Seattle, Washington
- Canada (8):
  - Regeneron Investigational Site, Calgary, Alberta
  - Regeneron Investigational Site, Surrey, British Columbia
  - Regeneron Investigational Site, Winnipeg, Manitoba
  - Regeneron Investigational Site, Markham, Ontario
  - Regeneron Investigational Site, Ottawa, Ontario
  - Regeneron Investigational Site, Peterborough, Ontario
  - Regeneron Research Site, Richmond Hill, Ontario
  - Regeneron Investigational Site, Windsor, Ontario

REFERENCES:
- [Derived] Langley RG, Gherardi G, Coleman A, Ardeleanu M, Rodriguez-Marco A, Levy S, Bansal A, Chen Z, Rossi AB, Shumel B, Khokhar FA. The Safety Data of Dupilumab for the Treatment of Moderate-to-Severe Atopic Dermatitis in Infants, Children, Adolescents, and Adults. Am J Clin Dermatol. 2025 Nov;26(6):981-1002. doi: 10.1007/s40257-025-00952-w. Epub 2025 Sep 24. PMID 40993471
- [Derived] Kamal MA, Kosloski MP, Lai CH, Partridge MA, Rajadhyaksha M, Kanamaluru V, Bansal A, Shabbir A, Shumel B, Ardeleanu M, Richards SM, Yan H, Xu CR, Rodriguez-Marco A, Xiao J, Khokhar FA, Gherardi G, Babilonia E, Maloney J, Mortensen E, Akinlade B, Braunstein N, Stahl N, Torri A, Davis JD, DiCioccio AT. Immunogenicity of dupilumab in adult and pediatric patients with atopic dermatitis. Front Immunol. 2024 Nov 11;15:1466372. doi: 10.3389/fimmu.2024.1466372. eCollection 2024. PMID 39588375
- [Derived] Paller AS, Silverberg JI, Cork MJ, Guttman-Yassky E, Lockshin B, Irvine AD, Kim MB, Kabashima K, Chen Z, Lu Y, Bansal A, Rossi AB, Shabbir A. Efficacy and Safety of Dupilumab in Patients With Erythrodermic Atopic Dermatitis: A Post Hoc Analysis of 6 Randomized Clinical Trials. JAMA Dermatol. 2023 Mar 1;159(3):255-266. doi: 10.1001/jamadermatol.2022.6192. PMID 36723913
- [Derived] Blauvelt A, Guttman-Yassky E, Paller AS, Simpson EL, Cork MJ, Weisman J, Browning J, Soong W, Sun X, Chen Z, Kosloski MP, Kamal MA, Delevry D, Chuang CC, O'Malley JT, Bansal A. Long-Term Efficacy and Safety of Dupilumab in Adolescents with Moderate-to-Severe Atopic Dermatitis: Results Through Week 52 from a Phase III Open-Label Extension Trial (LIBERTY AD PED-OLE). Am J Clin Dermatol. 2022 May;23(3):365-383. doi: 10.1007/s40257-022-00683-2. Epub 2022 May 14. PMID 35567671
- [Derived] Simpson EL, Paller AS, Siegfried EC, Thaci D, Wollenberg A, Cork MJ, Marcoux D, Huang R, Chen Z, Rossi AB, Shumel B, Sierka D, Bansal A. Dupilumab Demonstrates Rapid and Consistent Improvement in Extent and Signs of Atopic Dermatitis Across All Anatomical Regions in Pediatric Patients 6 Years of Age and Older. Dermatol Ther (Heidelb). 2021 Oct;11(5):1643-1656. doi: 10.1007/s13555-021-00568-y. Epub 2021 Aug 24. PMID 34427891
- [Derived] Kamal MA, Kovalenko P, Kosloski MP, Srinivasan K, Zhang Y, Rajadhyaksha M, Lai CH, Kanamaluru V, Xu C, Sun X, Simpson EL, Paller AS, Siegfried EC, Shumel B, Bansal A, Al-Huniti N, Davis JD. The Posology of Dupilumab in Pediatric Patients With Atopic Dermatitis. Clin Pharmacol Ther. 2021 Nov;110(5):1318-1328. doi: 10.1002/cpt.2366. Epub 2021 Aug 24. PMID 34270797
- [Derived] Siegfried EC, Bieber T, Simpson EL, Paller AS, Beck LA, Boguniewicz M, Schneider LC, Khokhar FA, Chen Z, Prescilla R, Mina-Osorio P, Bansal A. Effect of Dupilumab on Laboratory Parameters in Adolescents with Atopic Dermatitis: Results from a Randomized, Placebo-Controlled, Phase 3 Clinical Trial. Am J Clin Dermatol. 2021 Mar;22(2):243-255. doi: 10.1007/s40257-020-00583-3. Epub 2021 Mar 3. PMID 33655423
- [Derived] Bansal A, Simpson EL, Paller AS, Siegfried EC, Blauvelt A, de Bruin-Weller M, Corren J, Sher L, Guttman-Yassky E, Chen Z, Daizadeh N, Kamal MA, Shumel B, Mina-Osorio P, Mannent L, Patel N, Graham NMH, Khokhar FA, Ardeleanu M. Conjunctivitis in Dupilumab Clinical Trials for Adolescents with Atopic Dermatitis or Asthma. Am J Clin Dermatol. 2021 Jan;22(1):101-115. doi: 10.1007/s40257-020-00577-1. PMID 33481203
- [Derived] Silverberg JI, Yosipovitch G, Simpson EL, Kim BS, Wu JJ, Eckert L, Guillemin I, Chen Z, Ardeleanu M, Bansal A, Kaur M, Rossi AB, Graham NMH, Patel N, Gadkari A. Dupilumab treatment results in early and sustained improvements in itch in adolescents and adults with moderate to severe atopic dermatitis: Analysis of the randomized phase 3 studies SOLO 1 and SOLO 2, AD ADOL, and CHRONOS. J Am Acad Dermatol. 2020 Jun;82(6):1328-1336. doi: 10.1016/j.jaad.2020.02.060. Epub 2020 Mar 3. PMID 32135208
- [Derived] Paller AS, Bansal A, Simpson EL, Boguniewicz M, Blauvelt A, Siegfried EC, Guttman-Yassky E, Hultsch T, Chen Z, Mina-Osorio P, Lu Y, Rossi AB, He X, Kamal M, Graham NMH, Pirozzi G, Ruddy M, Eckert L, Gadkari A. Clinically Meaningful Responses to Dupilumab in Adolescents with Uncontrolled Moderate-to-Severe Atopic Dermatitis: Post-hoc Analyses from a Randomized Clinical Trial. Am J Clin Dermatol. 2020 Feb;21(1):119-131. doi: 10.1007/s40257-019-00478-y. PMID 31823222
- [Derived] Simpson EL, Paller AS, Siegfried EC, Boguniewicz M, Sher L, Gooderham MJ, Beck LA, Guttman-Yassky E, Pariser D, Blauvelt A, Weisman J, Lockshin B, Hultsch T, Zhang Q, Kamal MA, Davis JD, Akinlade B, Staudinger H, Hamilton JD, Graham NMH, Pirozzi G, Gadkari A, Eckert L, Stahl N, Yancopoulos GD, Ruddy M, Bansal A. Efficacy and Safety of Dupilumab in Adolescents With Uncontrolled Moderate to Severe Atopic Dermatitis: A Phase 3 Randomized Clinical Trial. JAMA Dermatol. 2020 Jan 1;156(1):44-56. doi: 10.1001/jamadermatol.2019.3336. PMID 31693077
- [Derived] Simpson EL, de Bruin-Weller M, Eckert L, Whalley D, Guillemin I, Reaney M, Chen Z, Nelson L, Qin S, Bansal A, Gadkari A. Responder Threshold for Patient-Oriented Eczema Measure (POEM) and Children's Dermatology Life Quality Index (CDLQI) in Adolescents with Atopic Dermatitis. Dermatol Ther (Heidelb). 2019 Dec;9(4):799-805. doi: 10.1007/s13555-019-00333-2. Epub 2019 Oct 22. PMID 31641952
- [Derived] Cork MJ, Thaci D, Eichenfield LF, Arkwright PD, Hultsch T, Davis JD, Zhang Y, Zhu X, Chen Z, Li M, Ardeleanu M, Teper A, Akinlade B, Gadkari A, Eckert L, Kamal MA, Ruddy M, Graham NMH, Pirozzi G, Stahl N, DiCioccio AT, Bansal A. Dupilumab in adolescents with uncontrolled moderate-to-severe atopic dermatitis: results from a phase IIa open-label trial and subsequent phase III open-label extension. Br J Dermatol. 2020 Jan;182(1):85-96. doi: 10.1111/bjd.18476. Epub 2019 Oct 8. PMID 31595499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 45 sites in the United States and Canada between 21 Mar 2017 and 05 Jun 2018. A total of 295 participants were screened, of which, 251 were eligible. The most common causes for screening failures were lack of adequate disease severity and lack of willingness to comply with study visits and procedures.
Pre-assignment Details: Eligible participants were randomized (1:1:1) & stratified by baseline Investigator's Global Assessment (IGA) score (3 vs 4) & body weight (<60 kg vs ≥60 kg) to 16 wks treatment with dupilumab every 2 wks (q2w) or q4w,or placebo q2w.
Groups:
- Placebo: Participants received placebo matching dupilumab once every 2 weeks (Q2W) (including doubling the amount of placebo on day 1 to match the loading dose). Participants in the <60-kilogram (kg) weight stratum received, in a 1:1 ratio, either placebo matching 200 milligram (mg) or placebo matching 300 milligram (mg). In the ≥60 kg weight stratum, the participants randomized to the placebo group received placebo matching 300 mg dupilumab.
- Dupilumab 300 mg Q4W: Participants received once every 4 weeks (Q4W) subcutaneous (SC) injections of 300 milligrams (mg) dupilumab following a loading dose of 600 mg on day 1. To maintain blinding, all participants received an injection once every 2 weeks (Q2W) from day 1 to week 14. Participants received placebo 2 millilitre (mL) injection at the weeks dupilumab was not given.
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Started | 85 | 84 | 82
Completed Wk 16 End of Treatment (EOT) | 80 | 81 | 79
Completed Week 28 (End of Study) | 2 | 4 | 3
Completed | 2 | 4 | 3
Not Completed | 83 | 80 | 79
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Lack of Efficacy | 3 | 1 | 0
Not completed — Discontinued to enroll in OLE: enrolled | 0 | 0 | 1
Not completed — Discont'd to enroll in OLE: not enrolled | 1 | 0 | 0
Not completed — Transitioned to OLE study | 76 | 76 | 73
Not completed — Withdrawal by Subject | 3 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W | Total
Number analyzed (Participants) | 85 | 84 | 82 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.78) | 14.4 (1.59) | 14.5 (1.74) | 14.5 (1.70)
Age, Customized [Number; unit: Participants]
  ≥12 to <15 years of age | 41 | 45 | 43 | 129
  ≥15 to <18 years of age | 44 | 39 | 39 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 39 | 103
  Male | 53 | 52 | 43 | 148
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 48 | 55 | 54 | 157
    Black or African American | 15 | 8 | 7 | 30
    Asian | 13 | 13 | 12 | 38
    Other | 6 | 8 | 7 | 21
    Not Reported/ Missing | 3 | 0 | 2 | 5
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity
  Participants
    Not Hispanic or Latino | 72 | 64 | 69 | 205
    Hispanic or Latino | 13 | 20 | 13 | 46
Duration of Atopic Dermatitis (AD) [Mean (Standard Deviation); unit: Years] | 12.3 (3.44) | 11.9 (3.18) | 12.5 (2.97) | 12.2 (3.20)
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: Scores on a scale] — The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
  Scores on a scale | 35.5 (13.97) | 35.8 (14.82) | 35.3 (13.84) | 35.5 (14.16)
Investigator's Global Assessment (IGA) Score [Count of Participants; unit: Participants] — IGA is an assessment scale used to determine severity of atopic dermatitis (AD) and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear).
  Participants
    IGA score = 3 (moderate) | 39 | 38 | 39 | 116
    IGA score = 4 (severe) | 46 | 46 | 43 | 135
Peak Weekly Averaged Pruritus Numerical Rating Scale (NRS) Score [Mean (Standard Deviation); unit: Peak weekly average score] — Peak Pruritus NRS is an assessment tool used by participants to report intensity of pruritus (itch) during a 24-hour recall period. Participants were asked the following question for maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable,' how would you rate your itch at the worst moment during the previous 24 hours?" Baseline NRS was the prorated average of NRSs reported continuously for 7 days right before and on the baseline visit (i.e., study day -6 to day 1).
  Peak weekly average score | 7.7 (1.62) | 7.5 (1.84) | 7.5 (1.52) | 7.6 (1.66)
Body Surface Area (BSA) of Atopic Dermatitis (AD) [Mean (Standard Deviation); unit: Percentage of BSA] — BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
  Percentage of BSA | 56.4 (24.13) | 56.9 (23.51) | 56.0 (21.40) | 56.5 (22.97)
Scoring Atopic Dermatitis (SCORAD) Score [Mean (Standard Deviation); unit: Scores on a scale] — The SCORAD index is a clinical tool for assessing the severity of atopic dermatitis. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
  Scores on a scale | 70.4 (13.25) | 69.8 (14.12) | 70.6 (13.89) | 70.3 (13.70)
Patient Oriented Eczema Measure (POEM) [Mean (Standard Deviation); unit: Scores on a scale] — The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in children and adults with atopic eczema. The format is participant response to 7 items (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) based on symptom frequency during the past week (ie, 0 = 'no days', 1 = '1 to 2 days', 2 = '3 to 4 days', 3 = '5 to 6' days, and 4 = 'every day'). The total score is the sum of the 7 items which is ranged from 0 to 28; a high score is indicative of a poor quality of life (QOL).
  Scores on a scale | 21.1 (5.38) | 21.1 (5.47) | 21.0 (5.01) | 21.0 (5.27)
Children's Dermatology Life Quality Index (CDLQI) Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The CDLQI is a 10-item questionnaire used to measure how much a participant's skin problem had affected the participant's quality of life (QOL) over a recall period of the past week. The questionnaire consists of 10 items. For each item the scale is rated as follows: 0 = Not at all = Not relevant; 1 = Only a little; 2 = Quite a lot; 3 = Very much = Yes = Prevents school. The CDLQI total score is the sum of the score of each question with a maximum of 30 and a minimum of 0. The higher the score, the greater the impact is on the QOL.
  Scores on a scale | 13.1 (6.72) | 14.8 (7.38) | 13.0 (6.21) | 13.6 (6.82)
Total Hospital Anxiety and Depression Scale (HADS) [Mean (Standard Deviation); unit: Scores on a scale] — The HADS is 14-item questionnaire with two subscales: anxiety & depression. Each item is rated on a 4-point scale (0-3). A person could score between 0 & 21 for each subscale (anxiety & depression). A high score is indicative of a poor state. Scores of 11 or more on either subscale are considered a 'definite case' of psychological morbidity, while scores of 8 to 10 represents 'probable case' & 0 to 7 'not a case'. The total score was the sum of the 2 sub-scores; therefore, the full range of possible values for the reported data is 0-42.
  Scores on a scale | 11.6 (7.76) | 13.3 (8.17) | 12.6 (8.04) | 12.5 (7.99)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) 0 or 1 (and Reduction From Baseline of ≥2 Points) at Week 16
Description: IGA is an assessment scale used to determine severity of atopic dermatitis (AD) and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). Participants with IGA "0" or "1" and a reduction from baseline of ≥2 points at Week 16 were reported. [Values after first rescue treatment used were set to missing. Participants with missing score at week 16 were considered as a non-responder. Participant considered non-responder after rescue treatment use. Efficacy analyses were based on the treatment allocated at randomization (as randomized).]
Time Frame: Baseline and Week 16
Population: Analysis was performed on Full Analysis Set (FAS) population (all randomized participants).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Percentage of participants | 2.4 | 17.9 | 24.4
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 200 mg or 300 mg Q2W; A hierarchical testing procedure was used to control type I error. Analysis was performed using Cochran-Mantel-Haenszel (CMH) test stratified by baseline disease severity (IGA=3 vs IGA=4) and baseline weight group (less than [<] 60 kilogram [kg] vs greater than or equal to [≥] 60 kg); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; percentage difference = 22, 95% CI 2-sided [12.2 to 31.87]
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg Q4W; A hierarchical testing procedure was used to control type I error. Analysis was performed using CMH test stratified by baseline disease severity (IGA=3 vs IGA=4) and baseline weight group (<60 kg vs ≥60 kg); Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; percentage difference = 15.5, 95% CI 2-sided [6.7 to 24.31]

2. Primary Outcome: Percentage of Participants With Eczema Area and Severity Index (EASI)-75 (≥75% Improvement From Baseline) at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI--75 responders were the participants who achieved ≥75% overall improvement in EASI score from baseline to Week 16. [Values after first rescue treatment used were set to missing. Participants with missing score at week 16 were considered as a non-responder. Participant considered nonresponder after rescue treatment use. Efficacy analyses were based on the treatment allocated at randomization (as randomized).]
Time Frame: Baseline and Week 16
Population: Analysis was performed on Full Analysis Set (FAS) population (all randomized participants).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Percentage of participants | 8.2 | 38.1 | 41.5
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 200 mg or 300 mg Q2W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; percentage difference = 33.2, 95% CI 2-sided [21.07 to 45.39]
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; percentage difference = 29.9, 95% CI 2-sided [17.94 to 41.78]

3. Secondary Outcome: Percent Change From Baseline in EASI Score at Week 16
Description: The Eczema Area and Severity Index (EASI) score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. [Values after first rescue treatment use were set to missing and participants with missing EASI score at Week 16 were considered as non-responders.]
Time Frame: Baseline and Week 16
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Percent change | -23.6 (5.49) [lower limit 5.49] | -64.8 (4.51) [lower limit 4.51] | -65.9 (3.99) [lower limit 3.99]
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 200 mg or 300 mg Q2W; A hierarchical testing procedure was used to control type I error. The confidence interval (CI) with p-value is based on treatment difference (Dupilumab group vs. Placebo) of the LS mean percent change using analysis of covariance (ANCOVA) model with baseline measurement as covariate and the treatment, randomization strata (baseline disease severity [IGA=3 vs IGA=4] and baseline weight group [<60 kg vs ≥60 kg]) as fixed factors; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; Least Square (LS) Mean difference = -42.3, 95% CI 2-sided [-55.6 to -29.04]
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg Q4W; A hierarchical testing procedure was used to control type I error. The confidence interval (CI) with p-value is based on treatment difference (Dupilumab group vs. Placebo) of the LS mean percent change using ANCOVA model with baseline measurement as covariate and the treatment, randomization strata (baseline disease severity [IGA=3 vs IGA=4] and baseline weight group [<60 kg vs ≥60 kg]) as fixed factors; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean difference = -41.2, 95% CI 2-sided [-54.44 to -28.02]

4. Secondary Outcome: Percent Change From Baseline in Weekly Average of Daily Peak Pruritus Numerical Rating Scale (NRS) Score at Week 16
Description: Peak Pruritus NRS is an assessment tool used by subjects to report intensity of pruritus (itch) during a 24-hour recall period. Participants were asked the following question: For maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable,' how would you rate your itch at the worst moment during the previous 24 hours?" For post-baseline NRS, the mean weekly NRS was calculated as the prorated average of the reported daily NRS within the week. For example, if there were 3 scores in a week, the prorated average = (score1 + score2 + score3) /3. [Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 16 were counted as non-responders.]
Time Frame: Baseline and Week 16
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Percent change | -19.0 (4.09) [lower limit 4.09] | -45.5 (3.54) [lower limit 3.54] | -47.9 (3.43) [lower limit 3.43]
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 200 mg or 300 mg Q2W; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean difference = -29, 95% CI 2-sided [-39.54 to -18.38]
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg Q4W; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean difference = -26.5, 95% CI 2-sided [-37.45 to 15.63]

5. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥3 Points) of Weekly Average of Daily Peak Pruritus NRS From Baseline to Week 16
Description: Peak Pruritus NRS is an assessment tool used by participants to report intensity of pruritus (itch) during a 24-hour recall period. Participants were asked the following question: For maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable,' how would you rate your itch at the worst moment during the previous 24 hours?" [For this endpoint, participants achieving a reduction of ≥3 points from baseline in weekly average of peak daily pruritus NRS score at Week 16 were reported. Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 16 were counted as non-responders.]
Time Frame: Baseline to Week 16
Population: Analysis was performed on FAS population (all randomized participants). Here, number of participants analyzed = participants with baseline peak pruritus NRS ≥3.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 83 | 82
Percentage of participants | 9.4 | 38.6 | 48.8
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 200 mg or 300 mg Q2W; A hierarchical testing procedure was used to control type I error. Difference is Dupilumab minus Placebo. C.I. = Confidence interval calculated using normal approximation. P-values were derived by CMH test stratified by baseline disease severity [IGA=3 vs IGA=4] and baseline weight group [<60 kg vs ≥60 kg]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; percentage difference = 39.4, 95% CI 2-sided [26.9 to 51.84]
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg Q4W; A hierarchical testing procedure was used to control type I error. Difference is Dupilumab minus Placebo. C.I. = Confidence interval calculated using normal approximation. P-values were derived by Cochran-Mantel-Haenszel (CMH) test stratified by baseline disease severity [IGA=3 vs IGA=4] and baseline weight group [<60 kg vs ≥60 kg]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; percentage difference = 29.1, 95% CI 2-sided [16.97 to 41.32]

6. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Weekly Average of Daily Peak Pruritus NRS From Baseline to Week 16
Description: Peak Pruritus NRS is an assessment tool used by participants to report intensity of pruritus (itch) during a 24-hour recall period. Participants were asked the following question: For maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable,' how would you rate your itch at the worst moment during the previous 24 hours?" [For this endpoint, participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 16 were reported. Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 16 were counted as non-responders.]
Time Frame: Baseline to Week 16
Population: Analysis was performed on FAS population (all randomized participants). Here, number of participants analyzed = participants with baseline peak pruritus NRS ≥4.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 84 | 83 | 82
Percentage of participants | 4.8 | 26.5 | 36.6
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 200 mg or 300 mg Q2W; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 31.8, 95% CI 2-sided [20.45 to 43.2]
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg Q4W; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 21.7, 95% CI 2-sided [11.21 to 32.28]

7. Secondary Outcome: Percentage of Participants With EASI-50 (≥50% Improvement From Baseline) at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-50 responders were the participants who achieved ≥50% overall improvement in EASI score at Week 16. [Values after first rescue treatment used were set to missing. Participants with missing value at Week 16 were considered as a non-responder].
Time Frame: Baseline and Week 16
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Percentage of participants | 12.9 | 54.8 | 61.0

8. Secondary Outcome: Percentage of Participants With EASI-90 (≥90% Improvement From Baseline) at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-90 responders were the participants who achieved ≥90% overall improvement in EASI score at Week 16. [Values after first rescue treatment used were set to missing. Participants with missing value at week 16 were considered as a non-responder.]
Time Frame: Baeline and Week 16
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Percentage of participants | 2.4 | 19.0 | 23.2

9. Secondary Outcome: Time to Onset of Effect on Pruritus as Measured by Percentage of Participants With Improvement (Reduction ≥3 Points) of Weekly Average of Daily Peak Pruritus NRS From Baseline
Description: as for outcome 5
Time Frame: Baseline up to week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 83 | 82
Percentage of participants | 11.4 (5.63) [lower limit 5.63] | 8.4 (5.92) [lower limit 5.92] | 7.7 (5.57) [lower limit 5.57]

10. Secondary Outcome: Time to Onset of Effect on Pruritus as Measured by Percentage of Participants With Improvement (Reduction ≥4 Points) of Weekly Average of Daily Peak Pruritus NRS From Baseline
Description: Peak Pruritus NRS is an assessment tool used by participants to report intensity of pruritus (itch) during a 24-hour recall period. Participants were asked the following question: For maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable,' how would you rate your itch at the worst moment during the previous 24 hours?" [For this endpoint, subjects achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 16 were reported. Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 16 were counted as non-responders.]
Time Frame: Baseline up to Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 84 | 83 | 82
Percentage of participants | 12.8 (4.90) [lower limit 4.90] | 9.9 (5.87) [lower limit 5.87] | 10.6 (5.50) [lower limit 5.50]

11. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) at Week 16
Description: BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
Time Frame: Baseline and Week 16
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Least Squares Mean (Standard Error); unit: Percentage of body surface area
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Percentage of body surface area | -11.66 (2.720) [lower limit 2.720] | -33.41 (2.330) [lower limit 2.330] | -30.11 (2.337) [lower limit 2.337]

12. Secondary Outcome: Percent Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Score at Week 16
Description: The SCORAD index is a clinical tool for assessing the severity of atopic dermatitis. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Time Frame: Baseline and Week 16
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Percent change | -17.6 (3.76) [lower limit 3.76] | -47.5 (3.21) [lower limit 3.21] | -51.6 (3.23) [lower limit 3.23]

13. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) Total Score at Week 16
Description: The CDLQI is a 10-item questionnaire used to measure how much a participant's skin problem had affected the participant's quality of life (QOL) over a recall period of the past week. The questionnaire consists of 10 items. For each item the scale is rated as follows: 0 = Not at all = Not relevant; 1 = Only a little; 2 = Quite a lot; 3 = Very much = Yes = Prevents school. The CDLQI total score is the sum of the score of each question with a maximum of 30 and a minimum of 0. The higher the score, the greater the impact is on the QOL.
Time Frame: Baseline and Week 16
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Scores on a scale | -5.1 (0.62) [lower limit 0.62] | -8.8 (0.53) [lower limit 0.53] | -8.5 (0.50) [lower limit 0.50]

14. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) at Week 16
Description: The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in children and adults with atopic eczema. The format is subject response to 7 items (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) based on symptom frequency during the past week (ie, 0 = 'no days', 1 = '1 to 2 days', 2 = '3 to 4 days', 3 = '5 to 6' days, and 4 = 'every day'). The total score is the sum of the 7 items which is ranged from 0 to 28; a high score is indicative of a poor quality of life (QOL).
Time Frame: Baseline and Week 16
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Scores on a scale | -3.8 (0.96) [lower limit 0.96] | -9.5 (0.86) [lower limit 0.86] | -10.1 (0.76) [lower limit 0.76]

15. Secondary Outcome: Change From Baseline in Weekly Average of Daily Peak Pruritus NRS at Week 16
Description: Peak Pruritus NRS is an assessment tool used by participants to report intensity of pruritus (itch) during a 24-hour recall period. Particpants were asked the following question for maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable,' how would you rate your itch at the worst moment during the previous 24 hours?" For post-baseline NRS, the mean weekly NRS was calculated as the prorated average of the reported daily NRS within the week. For example, if there were 3 scores in a week, the prorated average = (score1 + score2 + score3)/ 3.
Time Frame: Baseline and Week 16
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Scores on a scale | -1.54 (0.303) [lower limit 0.303] | -3.44 (0.260) [lower limit 0.260] | -3.70 (0.250) [lower limit 0.250]

16. Secondary Outcome: Percent Change From Baseline in Weekly Average of Daily Peak Pruritus NRS at Week 4
Description: Peak Pruritus NRS is an assessment tool used by participants to report intensity of pruritus (itch) during a 24-hour recall period. Participants were asked the following question for maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable,' how would you rate your itch at the worst moment during the previous 24 hours?" For post-baseline NRS, the mean weekly NRS was calculated as the prorated average of the reported daily NRS within the week. For example, if there were 3 scores in a week, the prorated average = (score1 + score2 + score3)/ 3.
Time Frame: Baseline and Week 4
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Percent change | -12.5 (3.06) [lower limit 3.06] | -33.1 (3.05) [lower limit 3.05] | -34.7 (2.99) [lower limit 2.99]

17. Secondary Outcome: Change From Baseline in Total Hospital Anxiety and Depression Scale (HADS) at Week 16
Description: The HADS is 14-item questionnaire with two subscales: anxiety & depression. Each item is rated on a 4-point scale (0-3). A person could score between 0 & 21 for each subscale (anxiety & depression). A high score is indicative of a poor state. Scores of 11 or more on either subscale are considered a 'definite case' of psychological morbidity, while scores of 8 to 10 represents 'probable case' & 0 to 7 'not a case'. The total score was the sum of the 2 sub-scores; therefore, the full range of possible values for the reported data is 0-42.
Time Frame: Baseline and Week 16
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Scores on a scale | -2.5 (0.80) [lower limit 0.80] | -5.2 (0.73) [lower limit 0.73] | -3.8 (0.68) [lower limit 0.68]

18. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Weekly Average of Daily Peak Pruritus NRS From Baseline at Week 4
Description: as for outcome 16
Time Frame: Baseline and Week 4
Population: Analysis was performed on FAS population (all randomized participants).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 84 | 82
Percentage of participants | 4.8 | 20.5 | 22.0

19. Secondary Outcome: Percentage of Participants With Skin-infection Treatment Emergent Adverse Events (TEAEs) (Excluding Herpetic Infections) Through Week 16
Description: Any untoward medical occurrence in a subject who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to the end of study (Week 16)). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline through Week 16
Population: Analysis was performed on FAS population (all randomized participants). Here, number of participants analyzed = participants with available data for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 83 | 82
Percentage of participants | 18.8 | 9.6 | 9.8

20. Secondary Outcome: Percentage of Participants With Serious TEAEs Through Week 16
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to the end of study (Week 28)). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline through Week 16
Population: as for outcome 19
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg Q2W
Number analyzed (Participants) | 85 | 83 | 82
Percentage of participants | 1.2 | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Day 197) regardless of seriousness or relationship to investigational product (IP).
Description: Of 251 participants randomized, 250 were included in Safety Analysis Set (SAF) reported here. (One participant in dupilumab Q4W arm was not dosed & was excluded from SAF). SAF analyzed as treated. Reported AEs are treatment-emergent AEs (TEAEs): developed/worsened during 'on treatment period' (from 1st dose of IP up to Day 113). TEAEs were collected for the 16-week treatment & follow-up period up to 12 weeks. After completing the treatment period, all were offered to enroll in study NCT02612454.
Groups:
- Dupilumab 200 mg or 300 mg: Participants with baseline weight <60 kg received once every 2 weeks (Q2W) subcutaneous (SC) injections of 200 milligrams (mg) dupilumab following a loading dose of 400 mg on day 1. Participants with baseline weight ≥60 kgreceived Q2W SC injections of 300 mg dupilumab following a loading dose of 600 mg on day 1.
Arm/Group | Placebo | Dupilumab 300 mg Q4W | Dupilumab 200 mg or 300 mg
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/83 | 0/82
Serious Adverse Events (participants affected / at risk) | 1/85 | 0/83 | 0/82
Other Adverse Events (participants affected / at risk) | 40/85 | 34/83 | 39/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=85) | Dupilumab 300 mg Q4W (N=83) | Dupilumab 200 mg or 300 mg (N=82)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=85) | Dupilumab 300 mg Q4W (N=83) | Dupilumab 200 mg or 300 mg (N=82)
Influenza (Infections and infestations) | 4 (4) | 0 (0) | 5 (6)
Nasopharyngitis (Infections and infestations) | 4 (5) | 10 (16) | 5 (8)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 5 (5) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 15 (23) | 7 (9) | 10 (13)
Headache (Nervous system disorders) | 9 (14) | 4 (5) | 9 (11)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 21 (29) | 16 (27) | 15 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT03054428/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT03054428/SAP_001.pdf